CLINICAL TRIAL: NCT01002924
Title: Protocol EC-FV-05: An Open-label, Multi-center, Extension Study of EC145 Administered Weeks 1 and 3 of a 4-Week Cycle in Subjects Enrolled in a Previous Study With EC145
Brief Title: Extension Study of EC145 (Vintafolide) for Subjects Enrolled in a Previous Study With EC145 (MK-8109-010)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8109-010; EC-FV-05
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumors
Keywords: Cancer; Adenocarcinoma; Phase II; Lung; Non-small cell lung cancer; NSCLC; extension; EC145; Prior exposure to EC145
MeSH Terms: conditions — Neoplasms; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — EC145

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participants invited to enroll on study will receive EC145 (vintafolide) 2.5 mg by intravenous bolus on Monday, Wednesday, and Friday of Weeks 1 and 3 in each 4-week cycle.
  Interventions: Drug: EC145

INTERVENTIONS:
Drug: EC145 — EC145 will be administered intravenously at a dose of 2.5 mg. Dosing will occur on Monday, Wednesday, and Friday of weeks 1 and 3 of each 4-week cycle. No therapy will be administered during weeks 2 and 4.

SUMMARY:
This extension protocol is for those subjects that have completed the allowed duration of participation in an Endocyte-sponsored clinical trial of EC145 (vintafolide) and have continuing evidence of clinical benefit (stable disease or better) at the time that they completed participation in that study.

DETAILED DESCRIPTION:
This extension protocol is for those subjects that have completed the allowed duration of participation in an Endocyte-sponsored clinical trial of EC145 and have continuing evidence of clinical benefit (stable disease or better) at the time that they completed participation in that study.

Following confirmation of eligibility, subjects will receive intravenously-administered EC145 at a dose of 2.5 mg. Dosing will occur on Monday, Wednesday, and Friday of weeks 1 and 3 of each 4-week cycle. No therapy will be administered during weeks 2 and 4. Subjects randomized to non-EC145-containing treatment arms of EC145 trials are not eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Must have received prior treatment with EC145 within the context of an Endocyte-sponsored, IRB-approved clinical trial.
* Disease (i.e., cancer) that was considered "stable" at the last evaluation while participating in the previous EC145-containing study. "Stable" is defined as not having progression of disease per standard criteria (RECIST, etc). Stable disease may be indicated by previously attained complete or partial tumor shrinkage that has not progressed per standard criteria.
* No more than 10 weeks have elapsed since the last evaluation of "stable disease".
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Must have recovered (to baseline/stabilization) from prior EC145-associated acute toxicities.
* Adequate bone marrow reserve, hepatic, and renal function.
* Negative serum pregnancy test for women of childbearing potential
* Willingness to practice contraceptive methods for men and women of childbearing potential.

Exclusion Criteria:

* Pregnancy.
* Development of a secondary malignancy requiring treatment.
* Symptomatic central nervous system (CNS) metastasis.
* History of receiving any investigational treatment or other systemic therapy directed at controlling cancer since the subject's last dose on the parent EC145 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-12-31 (Actual); Primary Completion 2013-12-11 (Actual); Study Completion 2013-12-11 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events | Up to 2 years
Number of participants experiencing serious adverse events | Up to 2 years
Number of participants discontinuing study drug due to adverse events | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Siu-Long Yao, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Center for Blood and Cancer Disorders, Bethesda, Maryland, United States